CLINICAL TRIAL: NCT04045912
Title: Reaching Adolescent Girls and Young Women Through Girl-Friendly Drug Vendors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); Health for a Prosperous Nation (Other); National Institute of Mental Health (NIMH) (NIH); Ministry of Health, Community Development, Gender, Elderly and Children, Tanzania (Unknown); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R34MH116804 (NIH); R34MH116804 (NIH)
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: HIV; Contraception
Keywords: HIV self-testing; Accredited drug dispensing outlets; Adolescent girls and young women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIVST + AGYW-Friendly Services (Experimental): Drug shops in Arm 1 will implement AGYW-friendly services, including a sexual and reproductive health (SRH) product display, a tablet with SRH videos, and a loyalty program ("the Queen Club") through which AGYW can earn mystery prizes and discreetly request free SRH products. They will also provide HIV self-test (HIVST) kits to AGYW customers for free.
  Interventions: Other: AGYW-Friendly Services; Other: HIVST
- HIVST Only (Active Comparator): Drug shops in Arm 2 will provide HIVST kits to AGYW customers for free.
  Interventions: Other: HIVST

INTERVENTIONS:
Other: AGYW-Friendly Services — Drug shops will offer a loyalty program (the "Queen Club") through which AGYW can earn mystery prizes and discreetly request free SRH products. Drug shops will also have an SRH product display and a tablet with SRH videos for interested customers, and drug shop employees will receive training on contraceptive counseling for AGYW.
  Arms: HIVST + AGYW-Friendly Services
Other: HIVST — Drug shops will provide HIVST kits to AGYW for free. Employees will receive training on HIVST and will institute an HIV care referral plan for customers who require linkage to confirmatory testing or treatment.

SUMMARY:
We will pilot an intervention to deliver sexual and reproductive health services, including HIV self-testing (HIVST) and contraception, to adolescent girls and young women (AGYW) at accredited drug dispensing outlets (ADDOs) in Shinyanga, Tanzania. In a 4-month randomized pilot study, we will compare mediating outcomes (AGYW patronage, product distribution, and referral) between 10 intervention and 10 comparison ADDOs, using data from time-location surveys of customers and inventory distribution and referral records.

DETAILED DESCRIPTION:
Building on our team's formative work using human-centered design methods and behavioral economics theories, we have designed an intervention (the "Queen Club") to develop AGYW-friendly drug shops where we will introduce HIVST alongside contraceptives and linkages to care. In a 4-month randomized pilot study, we will compare mediating outcomes (i.e., AGYW visits, distribution of HIVST and contraception, referral to SRH services) between 10 intervention and 10 comparison ADDOs, using data from a time-location survey of customers and records for HIVST and contraception distribution and referrals for sexual and reproductive health (SRH) services.

ADDOs will be randomly selected from four wards in the Shinyanga municipality. We will use stratified randomization by ward to assign 20 ADDOs 1:1 into the two study groups. Regardless of intervention arm, we will conduct the following activities in all ADDOs: in-person training on HIVST provision, monthly HIVST supply with half of kits explicitly earmarked for free provision to AGYW customers, an HIV care referral plan, and shop record tracking. The shop records will collect data on AGYW patronage, HIVST distribution, contraception distribution, and health facility referrals for SRH services. Monthly reviews of inventory records by the local team will include review of these records to determine AGYW patronage (for any service) and the volume and types of contraception and HIVST kits distributed to AGYW.

ADDOs in the intervention arm will be trained to implement the "Queen Club" intervention. The Queen Club intervention was developed through a year-long human-centered design process with AGYW and other stakeholders and is informed by behavioral economic theory and game-design. It is intended to partially mitigate to the physical, economic, and social constraints faced by AGYW in Shinyanga, as revealed in the formative research, and motivate them to discreetly seek HIVST and contraception at local drug shops, while in a context of fun.

In brief, the Queen Club is a loyalty program through which AGYW can earn surprise mystery gifts through repeated purchases at participating ADDOs. This is intended to build loyalty and trust with an ADDO shop, and also build the customer base for the ADDO owner. The back of the Queen Club loyalty card includes symbols, selected by AGYW, that represent oral contraception, HIVST, emergency contraception, condoms, and pregnancy tests. With the symbol portion of the card, AGYW can discreetly point to their desired product and receive it for free without questioning.

In a one-day training, we will review contraceptive methods and counseling techniques with intervention ADDO owners and staff using training materials adapted from the Ministry of Health, Community Development, Gender, Elderly, and Children. At every intervention ADDO, we will provide a countertop display with contraceptive methods and an HIVST kit for demonstration (if desired by any customer), as well as a tablet computer pre-loaded with videos about various contraceptive products and the Oraquick HIVST kit instructional video in Kiswahili.

The primary outcomes are mediators of the intervention's potential effect on preventing HIV and unintended pregnancy. In this phase, our goal is to measure these mediating, "process" outcomes and maximize learning for a future effectiveness and sustainability study using ADDOs as a platform to deliver HIVST and other HIV prevention and SRH services. We will collect data on the following mediating outcomes from the 10 intervention and 10 comparison ADDOs:

* AGYW patronage: number and proportion of visits by AGYW.
* Contraceptive distribution: number and types of contraceptives (i.e., condoms, oral contraception, emergency contraception) distributed to AGYW.
* Health facility referrals: number of referrals for AGYW made for SRH services, including HIV testing or treatment.
* HIVST kit uptake: number and proportion of kits distributed to AGYW.

We will assess AGYW patronage with a time-location survey of ADDO customers (randomly selected 3-hour intervals) at baseline (during the month prior to intervention) and during the final two months of the intervention (12 episodes per ADDO total) in which trained researchers will discreetly document the number of customers, their sex, and approximate age. Monthly reviews of inventory and referral records will show the volume and types of SRH products distributed to customers, including HIVST and contraception distributed to AGYW, and the number of SRH referrals made, the number and proportion for AGYW, and for which services.

We will compare AGYW patronage, referrals to health facilities, and contraception transactions between intervention and comparison ADDOs over the 4-month pilot period using: (1) statistical tests of means (t-tests) and medians (Wilcoxon rank-sum test); (2) a Poisson regression model (for counts of AGYW visits) to estimate rate ratios and confidence intervals controlling for baseline levels of AGYW patronage using a "difference-in-differences" approach; and (3) chi-squared tests for independence to qualitatively assess differences between groups for all mediating outcomes. Results will be used to understand the potential effectiveness of AGYW-friendly ADDO environments on AGYW visits and demand generation for HIV prevention and SRH services, a basis for power calculations to determine the sample size needed for the future study of effectiveness and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Owns an accredited drug dispensing outlet (ADDO);
* Willing to offer HIVST and AGYW-friendly services at drug shop;
* Provides written informed consent for the study.

Exclusion Criteria:

* Less than 18 years of age;
* Owns a drug shop that is not accredited;
* Unwilling to offer HIVST and/or AGYW-friendly services at drug shop;
* Does not provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Liu, PhD, MPP, MA, Principal Investigator — University of California, San Francisco
Locations (1):
- Health for a Prosperous Nation, Shinyanga, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willard-Grace R, Abigail Cabrera F, Bykhovsky C, Douglas K, Hunter LA, Mnyippembe A, Mgunya KH, McCoy SI, Liu JX. "They call me the 'Great Queen'": implementing the Malkia Klabu program to improve access to HIV self-testing and contraception for adolescent girls and young women in Tanzania. Reprod Health. 2024 Feb 7;21(1):21. doi: 10.1186/s12978-024-01744-x. PMID 38321482
- [Derived] Hunter LA, Rao A, Napierala S, Kalinjila A, Mnyippembe A, Hassan K, Bertozzi SM, Mfaume R, Njau P, Liu JX, McCoy SI. Reaching Adolescent Girls and Young Women With HIV Self-Testing and Contraception at Girl-Friendly Drug Shops: A Randomized Trial in Tanzania. J Adolesc Health. 2023 Jan;72(1):64-72. doi: 10.1016/j.jadohealth.2022.08.013. Epub 2022 Oct 12. PMID 36241492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We randomly selected 41 drug shops from a registry of Accredited Drug Dispensing Outlets that included contact information for the shops' primary shopkeepers. Of the 41 shopkeepers, 14 were ineligible and 6 could not be contacted. Of the 21 shopkeepers that were eligible and could be contacted, 20 consented to participate (corresponding to 20 participating drug shops). Adolescent girls and young women (AGYW) customers were not enrolled as participants in this trial.
Pre-assignment Details: Enrollment and pre-randomization baseline data collection began July 22, 2019 and ended August 17, 2019. All participating drug shopkeepers were randomized into study arms on August 19, 2019.
Units Other Than Participants: drug shops
Groups:
- HIVST + AGYW-Friendly Services: Drug shops in Arm 1 will implement adolescent girl and young women (AGYW)-friendly services, including a sexual and reproductive health (SRH) product display, a tablet with SRH videos, and a loyalty program ("the Queen Club") through which AGYW can earn mystery prizes and discreetly request free SRH products. They will also provide HIV self-test (HIVST) kits to AGYW customers for free.
  AGYW-Friendly Services: Drug shops will offer a loyalty program (the "Queen Club") through which AGYW can earn mystery prizes and discreetly request free SRH products. Drug shops will also have an SRH product display and a tablet with SRH videos for interested customers, and drug shop employees will receive training on contraceptive counseling for AGYW.
  HIVST: Drug shops will provide HIVST kits to AGYW for free. Employees will receive training on HIVST and will institute an HIV care referral plan for customers who require linkage to confirmatory testing or treatment.
- HIVST Only: Drug shops in Arm 2 will provide HIV self-test (HIVST) kits to adolescent girl and young women (AGYW) customers for free.
  HIVST: Drug shops will provide HIVST kits to AGYW for free. Employees will receive training on HIVST and will institute an HIV care referral plan for customers who require linkage to confirmatory testing or treatment.
Period: Overall Study
Arm/Group | HIVST + AGYW-Friendly Services | HIVST Only
Started | 10; 10 drug shops | 10; 10 drug shops
Completed | 10; 10 drug shops | 10; 10 drug shops
Not Completed | 0; 0 drug shops | 0; 0 drug shops

BASELINE CHARACTERISTICS:
Units Other Than Participants: drug shops
Groups:
- Total: Total of all reporting groups
Arm/Group | HIVST + AGYW-Friendly Services | HIVST Only | Total
Number analyzed (Participants) | 10 | 10 | 20
Number analyzed (drug shops) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (15.3) | 38.7 (15.7) | 43.6 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 10 | 10 | 20
Location of drug shop [Count of Units; unit: drug shops]
  Ward 1 | 3 | 3 | 6
  Ward 2 | 3 | 3 | 6
  Ward 3 | 2 | 2 | 4
  Ward 4 | 2 | 2 | 4
Number of people who work in drug shop [Count of Units; unit: drug shops]
  1 person | 7 | 10 | 17
  2 people | 2 | 0 | 2
  3 people | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: AGYW Patronage (Count)
Description: Number of visits by adolescent girls and young women (AGYW) during drug shop observations at baseline (before randomization), midline (after 2-3 months), and endline (after 3-4 months).
Time Frame: Baseline (pre-randomization) through Month 4
Population: We randomly sampled five 3-hour observation day/time blocks per shop per time point, corresponding to up to 15 observations per shop across the study period.
Measure: Mean (Standard Deviation); unit: AGYW customers per observation
Units Other Than Participants: drug shop observations
Arm/Group | HIVST + AGYW-Friendly Services | HIVST Only
Number analyzed (Participants) | 10 | 10
Number analyzed (drug shop observations) | 141 | 132
AGYW customers per observation
  Baseline (pre-randomization): number analyzed (drug shop observations) | 45 | 40
  Baseline (pre-randomization) | 1.0 (1.2) | 1.0 (1.1)
  Midline: number analyzed (drug shop observations) | 47 | 44
  Midline | 1.7 (2.9) | 1.0 (1.3)
  Endline: number analyzed (drug shop observations) | 49 | 48
  Endline | 4.0 (5.2) | 0.8 (1.2)
  Midline/endline combined: number analyzed (drug shop observations) | 96 | 92
  Midline/endline combined | 2.9 (4.4) | 0.9 (1.2)

2. Primary Outcome: AGYW Patronage (Proportion)
Description: Proportion of visits by AGYW during drug shop observations at baseline (before randomization), midline (after 2-3 months), and endline (after 3-4 months); calculated as the number of AGYW customers divided by the total number of customers per observation.
Time Frame: Baseline (pre-randomization) through Month 4
Population: We randomly sampled five 3-hour observation day/time blocks per shop per time point, corresponding to up to 15 observations per shop across the study period. Unlike the first AGYW patronage outcome, this outcome excludes observations during which zero customers were observed.
Measure: Mean (Standard Deviation); unit: Proportion of AGYW customers
Units Other Than Participants: drug shop observations
Arm/Group | HIVST + AGYW-Friendly Services | HIVST Only
Number analyzed (Participants) | 10 | 10
Number analyzed (drug shop observations) | 134 | 127
Proportion of AGYW customers
  Baseline (pre-randomization): number analyzed (drug shop observations) | 42 | 40
  Baseline (pre-randomization) | 0.17 (0.19) | 0.12 (0.13)
  Midline: number analyzed (drug shop observations) | 43 | 41
  Midline | 0.22 (0.28) | 0.12 (0.12)
  Endline: number analyzed (drug shop observations) | 49 | 46
  Endline | 0.39 (0.31) | 0.11 (0.21)
  Midline/endline combined: number analyzed (drug shop observations) | 92 | 87
  Midline/endline combined | 0.31 (0.31) | 0.12 (0.17)

3. Primary Outcome: HIVST Kit Uptake
Description: Number of HIV self-test (HIVST) kits distributed to AGYW over four months of post-randomization study arm implementation. Drug shopkeepers maintained standardized records of the number of HIVST kits distributed to AGYW customers in participating drug shops throughout the implementation period.
Time Frame: Month 1 (post-randomization) through Month 4
Measure: Mean (Standard Deviation); unit: HIVST kits distributed per shop
Units Other Than Participants: drug shops
Arm/Group | HIVST + AGYW-Friendly Services | HIVST Only
Number analyzed (Participants) | 10 | 10
Number analyzed (drug shops) | 10 | 10
HIVST kits distributed per shop | 145.6 (107.6) | 59.6 (30.4)

4. Primary Outcome: Contraceptive Distribution
Description: Number of contraceptives distributed to AGYW, including condoms, oral contraception, and emergency contraception, over four months of post-randomization study arm implementation. Drug shopkeepers maintained standardized records of the number and types of contraceptives distributed to AGYW customers in participating drug shops throughout the implementation period.
Time Frame: Month 1 (post-randomization) through Month 4
Measure: Mean (Standard Deviation); unit: Contraceptives provided per shop
Units Other Than Participants: drug shops
Arm/Group | HIVST + AGYW-Friendly Services | HIVST Only
Number analyzed (Participants) | 10 | 10
Number analyzed (drug shops) | 10 | 10
Contraceptives provided per shop
  Contraceptives (all) | 664.9 (1073.5) | 19.9 (27.4)
  Condoms | 128.9 (142.7) | 12.3 (25.8)
  Daily oral contraception | 77.3 (60.5) | 3.6 (5.3)
  Emergency contraception | 458.7 (904.4) | 4.0 (4.9)

5. Primary Outcome: Health Facility Referrals
Description: Number of health facility referrals provided to AGYW for sexual and reproductive health (SRH) services, including HIV testing/treatment, family planning, and pregnancy services, over four months of post-randomization study arm implementation. Drug shopkeepers maintained standardized records of the number and types of SRH health facility referrals provided to AGYW customers in participating drug shops throughout the implementation period.
Time Frame: Month 1 (post-randomization) through Month 4
Measure: Mean (Standard Deviation); unit: Referrals provided per shop
Units Other Than Participants: drug shops
Arm/Group | HIVST + AGYW-Friendly Services | HIVST Only
Number analyzed (Participants) | 10 | 10
Number analyzed (drug shops) | 10 | 10
Referrals provided per shop
  SRH referrals (all) | 66.1 (157.5) | 6.7 (19.1)
  HIV referrals | 8.2 (20.0) | 0.2 (0.4)
  Family planning referrals | 49.5 (120.0) | 4.9 (15.1)
  Pregnancy referrals | 8.4 (17.8) | 1.6 (4.0)

6. Secondary Outcome: Pregnancy Test Distribution
Description: Number of urine pregnancy tests distributed to AGYW over four months of post-randomization study arm implementation. Drug shopkeepers maintained standardized records of the number of pregnancy tests distributed to AGYW customers in participating drug shops throughout the implementation period.
Time Frame: Month 1 (post-randomization) through Month 4
Measure: Mean (Standard Deviation); unit: Pregnancy tests provided per shop
Units Other Than Participants: drug shops
Arm/Group | HIVST + AGYW-Friendly Services | HIVST Only
Number analyzed (Participants) | 10 | 10
Number analyzed (drug shops) | 10 | 10
Pregnancy tests provided per shop | 182.2 (236.0) | 28.1 (29.0)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Shopkeepers were encouraged to contact the research team if any adverse events occurred. Research assistants also asked about adverse events as part of study close-out procedures.
Arm/Group | HIVST + AGYW-Friendly Services | HIVST Only
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
This pilot trial included 10 intervention shops, all located within the specific context in which the intervention was designed. Future studies are needed to evaluate the intervention in other settings. Research assistants conducting shop observations and shopkeepers completing customer logs relied on visual assessment of customer age. There may be measurement error associated with the use of shopkeepers' logs to assess the distribution of SRH products and health facility referrals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT04045912/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT04045912/ICF_001.pdf